CLINICAL TRIAL: NCT05720676
Title: Clinical, Histopathological, Molecular and Experimental Characterization of Liver Metastases From Patients With Breast Cancer.
Brief Title: Clinical, Histological and In-depth Molecular Characterization as Well as Experimental Models of Liver Metastasis From Patients With Breast Cancer in Order to Identify New Potential Treatment Avenues.
Acronym: OLiver Pro
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Collaborators: Jules Bordet Institute (Other); Erasme University Hospital (Other); GZA Ziekenhuizen Campus Sint-Augustinus (Other)
Responsible Party: Principal Investigator, Sophia Leduc, PhD Student, KU Leuven
Other Study IDs: S-64813
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Liver Metastases
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about breast cancer liver metastasis in patients who met the following criteria:

* female;
* be ≥ 18 years of age on the day of signing informed consent;
* confirmed diagnosis of breast cancer liver metastases. Newly diagnosed patients with de-novo liver metastases are eligible;
* be planned for liver surgery.

The main questions it aims to answer are:

1. To characterize the tumour cells and their microenvironment in the liver metastases at the transcriptomic and protein single-cell level;
2. To determine the levels and patterns of immune infiltrates in liver metastases from BC patients;
3. To identify biological features associated with the histopathological growth patterns in liver metastases.
4. To create patient-derived xenografts (PDX) and organoids (PDO) from liver metastases isolated from patients with BC;
5. To perform a histopathological and molecular comparison of liver metastases, PDX and PDO isolated from the same patient

Participants will be willing and able to provide written informed consent for this study and tissue samples for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* be willing and able to provide written informed consent for this study;
* female;
* be ≥ 18 years of age on the day of signing informed consent;
* confirmed diagnosis of breast cancer liver metastases. Newly diagnosed patients with de-novo liver metastases are eligible;
* be planned for liver surgery;
* be willing to provide tissue samples for research purposes.

Exclusion Criteria:

* unwillingness to provide the samples or clinical information needed for the study;
* History of radiofrequency destruction (RF), stereotactic Body Radiotherapy (SBRT) or intra-arterial treatment such as chemoembolization (TACE) or selective internal radiation therapy (SIRT) performed on the metastasis to be examined (accepted if performed in other metastasis);
* Has an active autoimmune disease that has required systemic treatment in the past 2 years prior to the surgery (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment;
* Presence of immunodeficiency or immune dysregulatory diseases and conditions which require active immune modulatory treatment of any kind, or required treatment in the past two years from date of diagnosis of breast cancer;
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results in the opinion of the treating investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who are planned for liver surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
To characterize the tumour cells and their microenvironment in the liver metastases at the transcriptomic and protein single-cell level. | 2 years
To determine the levels and patterns of immune infiltrates in liver metastases from BC patients | 2 years
To identify biological features associated with the histopathological growth patterns in liver metastases. | 2 years
To create patient-derived xenografts (PDX) and organoids (PDO) from liver metastases isolated from patients with BC | 2 years
To perform a histopathological and molecular comparison of liver metastases, PDX and PDO isolated from the same patient. | 2 years
To investigate the histopathological growth patterns of liver metastases using intra-vital imaging of these metastases in PDX. | 2 years
To use PDX and PDO to evaluate the efficacy of various treatments. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sophia Leduc, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided